CLINICAL TRIAL: NCT00003588
Title: A Phase I Study of Ad-p53 (NSC# 683550) for Patients With Platinum- and Paclitaxel-Resistant Epithelial Ovarian Cancer
Brief Title: Gene Therapy in Treating Patients With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02277; MDA-ID-97228; NCI-T97-0111; CDR0000066657 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2002-06

CONDITIONS: Ovarian Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — advexin; Laparoscopy

ARMS (1):
- Arm I (Experimental): Patients undergo laparoscopy for p53 assessment and catheter placement. Patients receive daily intraperitoneal injections of adenovirus p53 (Ad-p53) for 5 days every 3 weeks. Treatment is repeated every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients each are treated at each dose level of Ad-p53. The maximum tolerated dose is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity.
  Interventions: Biological: Ad5CMV-p53 gene; Procedure: laparoscopic surgery

INTERVENTIONS:
Biological: Ad5CMV-p53 gene
Procedure: laparoscopic surgery

SUMMARY:
Phase I trial to study the effectiveness of gene therapy in treating patients with ovarian cancer that has not responded to previous treatment. Inserting the p53 gene into a person's cancer cells may improve the body's ability to fight cancer or make the cancer cells more sensitive to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated doses of adenovirus p53 in patients with platinum- and paclitaxel-resistant ovarian epithelial cancer.

II. Determine the qualitative and quantitative toxic effects of this regimen in these patients.

III. Document the observed anti-tumor activity of this regimen in these patients.

IV. Evaluate the biological endpoints (e.g., induction of apoptosis, p53 expression) of this regimen in these patients.

OUTLINE: This is a dose escalation study.

Patients undergo laparoscopy for p53 assessment and catheter placement. Patients receive daily intraperitoneal injections of adenovirus p53 (Ad-p53) for 5 days every 3 weeks. Treatment is repeated every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients each are treated at each dose level of Ad-p53. The maximum tolerated dose is defined as the dose at which no more than 1 of 6 patients experiences dose limiting toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic ovarian epithelial cancer that is platinum- and paclitaxel resistant as defined by: Disease progression while on first-line regimen containing both a platinum drug and paclitaxel OR Tumor progression within 6 months of completion of platinum-based therapy (either as first- or second-line) or paclitaxel-based therapy (either as first- or second-line)
* Refractory or recurrent ovarian epithelial cancer as defined by: Lesions of any diameter
* Nonmeasurable disease (with CA-125 at least 35)
* Ascites and/or pleural effusions allowed
* No borderline or low malignant potential tumors

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: Zubrod 0-2
* Life expectancy: At least 12 weeks
* WBC at least 3,000/mm3
* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.5 mg/dL PT/PTT normal
* Creatinine no greater than 1.4 mg/dL
* No active, unresolved upper respiratory infections
* Not HIV positive
* At least 5 years since prior malignancy, except nonmelanomatous skin cancer
* Willing and able to undergo placement of Tenckhoff catheter in the peritoneal cavity for sampling of ascites or peritoneal fluid
* No concurrent serious medical illness
* No untreated gastrointestinal obstruction
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* May have failed an unlimited number of prior chemotherapy regimens
* At least 30 days since prior chemotherapy
* No prior radiotherapy to the pelvis or abdomen
* Eligible for laparoscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1998-09; Primary Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith K. Wolf, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States